CLINICAL TRIAL: NCT04946643
Title: Contribution of Subclavian Vein Diameter Variations to Assess Vascular Filling Among Critical Care Patients
Brief Title: Subclavian Vein Diameter Variations to Assess Vascular Filling
Acronym: VSC MIR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210513; 2021-A00694-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-06-21; First posted 2021-07-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Circulatory Failure
Keywords: acute circulatory failure; intensive care unit; echocardiography; superior and inferior vena cava
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Haemodynamic optimisation is a fundamental step and a daily issue in the management of intensive care patients with acute circulatory failure. Failure to optimise haemodynamics is recognised as a factor associated with morbidity and mortality.

Although the first line of treatment is often vascular filling, many studies have found that excessive vascular filling alone is deleterious and leads to increased morbidity and mortality due to pulmonary and interstitial oedema. The use of catecholamines avoids this undue vascular filling.

At present, the therapeutic strategy in acute circulatory failure is to perform a personalised "titrated" vascular filling after assessing the need for it.

To do this, predictive criteria for the need to continue vascular filling in order to optimise cardiac output and tissue perfusion pressure, particularly by ultrasound, have been developed, notably by transesophageal approach.

It also appeared to us that offering an alternative to the transesophageal approach would reduce invasiveness on the one hand, but would also offer an alternative when the transesophageal approach is contraindicated.

DETAILED DESCRIPTION:
Acute circulatory failure is encountered in shock, regardless of its origin, when physiological compensatory mechanisms are overwhelmed. The initial tachycardia and reflex vasoconstriction of shock aims to maintain sufficient arterial pressure and tissue perfusion pressure. Beyond these mechanisms of compensation for relative and/or absolute hypovolaemia, arterial hypotension and tissue hypoperfusion appear, expressed clinically by functional signs (e.g. asthenia) and physical signs (arterial hypotension, consciousness disorders, mottling, oliguria, etc.).

It has been observed that organ failure induced by circulatory insufficiency is associated with a poor prognosis in septic shock. In daily clinical practice, acute circulatory failure is most often characterised by haemodynamic failure as reflected by arterial hypotension and/or tachycardia. Early treatment of acute circulatory failure is a recognised prognostic factor in trauma patients and patients with septic shock (2,3), leading to a reduction in mortality.

The first line of treatment for circulatory failure is usually early vascular filling due to relative and absolute hypovolaemia. The choice of fluids depends on the clinical situation, although for septic shock crystalloids are recommended as first-line therapy. Although early vascular filling is the first line of treatment, overfilling, also known as "induced" vascular filling, is alone recognised as a factor associated with excess mortality in various situations of acute circulatory failure. It is now accepted that early administration of inotropic and/or vasopressor agents, i.e. before the end of vascular filling, is necessary to restore arterial pressure and therefore limit the consequences of tissue hypo perfusion. In order to determine the choice between continued vascular filling and the administration of vasopressor and/or inotropic agents, predictive indicators of vascular filling requirements have been developed. These aim to determine whether or not vascular filling will increase cardiac output or one of its surrogates such as the subaortic time velocity integral (SATI).

Numerous indicators have been described for more than 30 years in intensive care units. Dynamic criteria are those that have the best predictive performance compared to static indicators. Their time-consuming implementation requires an invasive approach for most of these criteria due to their technical nature and the need to respect sometimes restrictive validity criteria.

The technological development of ultrasound scanners has allowed their liberal use and the validation of dynamic ultrasound criteria predictive of the response to vascular filling (respiratory variations of the sub-aortic velocity time integral, S wave, index of distensibility of the inferior vena cava, index of collapsibility of the superior vena cava, central venous pressure). The mechanism underlying superior vena cava collapsibility is complex, involving variations in intra-thoracic pressure as well as the inherent movements of the lung parenchyma. These pathophysiological mechanisms have not yet been described.

A recent study has demonstrated the interchangeability between delta PP and respiratory variations in subclavian vein diameter in intensive care patients and in the operating theatre.

The advantages of the transthoracic ultrasound approach to assessing respiratory variations in subclavian vein diameter are its rapidity of implementation, ease of use, non-invasive nature and reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Acute circulatory failure from any cause defined as low blood pressure (systolic blood pressure less than 90mmHg and/or mean arterial pressure less than 65mmHg) and/or marbling and mechanical ventilation;
* Affiliation with a social security scheme or entitled to it;
* Information and non-objection of the patient to participate in the research.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age over 18 years, Acute circulatory failure from any cause defined as low blood pressure (systolic blood pressure less than 90mmHg and/or mean arterial pressure less than 65mmHg) and/or marbling and mechanical ventilation, affiliation with a social security scheme or entitled to it, information and non-objection of the patient to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Respiratory variations of subclavian vein diameter | at 5 minutes
  Correlation between respiratory variations in subclavian vein (SCV) diameter with cardiac output assessed by measuring respiratory variations in the subaortic velocity time integral

SECONDARY OUTCOMES:
Collapsibility index of the superior vena cava | at 5 minutes
  Correlation between respiratory variations in subclavian vein (SCV) diameter and collapsibility index of the superior vena cava assessed by trans thoracic and trans oesophageal approach.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, PhD, Principal Investigator — Intensive care unit, Ambroise Paré hospital, APHP
Locations (1):
- Intensive care unit, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No